CLINICAL TRIAL: NCT02799524
Title: Comparison of Mood Disorders Screening Scales in Geriatric Oncology
Acronym: Thymog
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Collaborators: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-A00836-43; 15-087 (Other: CHU Caen)
Record Dates: First submitted 2016-04-01; First posted 2016-06-15 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-01

CONDITIONS: Mood Disorders
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: comparison of screening scales — Concordance degrees Assessment of each of 2 scales ( HADS and GDS ) from the DSM- V , for diagnostic confirmation of major depressive episodes in elderly patients with cancer or haematological malignancies

SUMMARY:
The objective of this study is to evaluate the scales commonly used in geriatrics and oncology distress thermometer ( analogue scale rated from 0 to 1 for the emotional distress ) , the GDS15 (15 issues closed binary response seeking signs of depression ) the HADS (14 questions assessing the intensity of anxiety signs and signs of depression listed 0-3 ).

The prospective observational study will be conducted in parallel on two sites ( University Hospital Centre and François Baclesse ) after informed patient information.

It will be offered to patients 70 years and over with a new diagnosis or relapse of cancer or haematological malignancies in the hospital to meet the mood disorder screening questionnaires .

DETAILED DESCRIPTION:
There are various tools validated and recommended by the SiO and SFPO for screening mood disorders in geriatric oncology . The choice among them depends on the usual practices of the various teams , only some scales assessing depressive signs and other signs of anxiety too. None were assessed in a population aged diagnosis of cancer or hematologic malignancy in pre- therapeutic situation.

The objective of this study is to evaluate the scales commonly used in geriatrics and oncology distress thermometer ( analogue scale rated from 0 to 1 for the emotional distress ) , the GDS15 (15 issues closed binary response seeking signs of depression ) the HADS (14 questions assessing the intensity of anxiety signs and signs of depression listed 0-3 ) The prospective observational study will be conducted in parallel on two sites ( University Hospital Centre and François Baclesse ) after informed patient information.

It will be offered to patients 70 years and over with a new diagnosis or relapse of cancer or haematological malignancies in the hospital to meet the mood disorder screening questionnaires .

If one test is abnormal , a clinical psychological care will be offered . When returning home : telephone contact will be made the same day with the doctor , asking him to please make thymic revaluation within 2 weeks ( informed patient). It will be sent to the doctor by post a rubric of Major Depressive Episode criteria of the DSM V to return . If the patient remains hospitalized , the doctor taking care of patient will be contacted to obtain the same information .

In addition, the investigators will study the impact on the management (change or introduction of an antidepressant and / or anxiolytic use of psychotherapy or psychological counseling ... ) to 5 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patient 70 years and older with diagnosis of cancer or haematological malignancies ,
* New diagnosis or relapse announced
* Supported in the 2 c among : in consultation , or hospital geriatric or oncology / hematology specialty
* Affiliated Health Insurance

Exclusion Criteria:

* Cognitive problems preventing self

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Men and women 70 years and older with newly diagnosed or relapsed cancer or haematological malignancies (not older than one month)
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Concordance degrees Assessment (HADS and GDS ) | 3 weeks
  Concordance degrees Assessment of each of 2 scales ( HADS and GDS ) from the DSM- V , for diagnostic confirmation of major depressive episodes in elderly patients with cancer or haematological malignancies

SECONDARY OUTCOMES:
Correlation between the presence of signs of depression screening by HADS -D ( ≥11 / 21) and GDS ( > 5/15) | 3 weeks
  Correlation between the presence of signs of depression screening by HADS -D ( ≥11 / 21) and GDS ( > 5/15) with the following factors: the type of cancer, concept of relapse, there is an oncologic therapeutic project or no , sex , social status, loss of autonomy, presence of pain , severe comorbidities ( CIRS - G≥3 ) , psychiatric history , psychotropic treatment ( anxiolytic , antidepressant) in place
correlation between anxious signs of HADS -A ( ≥11 / 21) and the distress thermometer ( ≥4 / 10) and factors outcome 2 | 3 weeks
  correlation between anxious signs of HADS -A ( ≥11 / 21) and the distress thermometer ( ≥4 / 10) and the type of cancer, concept of relapse, oncologic therapeutic project or no, sex, social status, loss of autonomy, presence of pain, severe comorbidities, psychiatric history , psychotropic treatment in place
Comparison of the distress thermometer score between screening and revaluation to 3 weeks | 3 weeks
  Comparison of the distress thermometer score between screening and revaluation to 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Caen UH, Caen, France

IPD SHARING:
Plan to Share IPD: No